CLINICAL TRIAL: NCT04903808
Title: Clinical And Cost- Effectiveness of Allium Sativum Oil Versus Mineral Trioxide Aggregate in Primary Molars Pulpotomy in Group of Egyptian Children : A Randomised Clinical Pilot Study.
Brief Title: Clinical And Cost- Effectiveness of Allium Sativum Oil (Garlic Oil ) Versus Mineral Trioxide Aggregate in Primary Molars Pulpotomy in Group of Egyptian Children : A Randomised Clinical Pilot Study.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lobna Magdy, Researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lobnamagdy128
Record Dates: First submitted 2021-05-20; First posted 2021-05-27 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Carious Primary Molars
Keywords: Allium sativum oil; MTA; pulpotomy
MeSH Terms: interventions — allyl sulfide; TheraCal; Pemetrexed

STUDY DESIGN:
Intervention Model Description: It is a double-blinded randomised clinical trial with equal randomisation parallel design with allocation ratio 1:1
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and outcome assessor will be blinded (double blind study )
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allium sativum oil (Experimental): The pulp stumps of the molars are dressed with a cotton pellet that is made damp with Allium Sativum oil for 1 min .
  Interventions: Drug: Allium Sativum Oil
- Mineral Trioxide Aggregate (Active Comparator): The material will be prepared according to the manufacturer's instructions , applied to the pulp chamber and a moistened cotton pellet was placed over the MTA paste to allow the material to set.
  Interventions: Drug: Mineral Tri-Oxide Aggregate

INTERVENTIONS:
Drug: Allium Sativum Oil — Garlic oil Captain Company (CAP-PHARM)
  Other Names: Garlic oil
  Arms: Allium sativum oil
Drug: Mineral Tri-Oxide Aggregate — ProRoot MTA, Dentsply
  Other Names: MTA
  Arms: Mineral Trioxide Aggregate

SUMMARY:
Allium Sativum oil is advocated to prove the capability of new natural products in replacing higher cost pharmacological materials, while achieving the same successful clinical and radiographic long-term results.

DETAILED DESCRIPTION:
One of the most challenging subjects in paediatric dentistry is choosing the ideal pulp medication material that has the required properties such as preserving the vitality of the remaining intact pulp and stimulating its repair. This material should prevent pathological root resorption.Clinical and cost effectiveness trials from different countries are useful to determine which medicament should be advocated in which economic setting . Alternative pulpotomy materials clinically effective as MTA but with lower cost should be studied .

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy children aged from 5- 7 years.
* Children not having antibiotics in the past 14 days.
* Cooperative children.
* Children are having at least two carious asymptomatic second primary molars.

Exclusion Criteria:

* Uncooperative children.
* Immunocompromised children.
* Children with clinical or radiographic symptoms

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Clinical effectiveness | 1 year follow up
  clinical effectiveness will be measured by intraoral examination and radiographic assessment

SECONDARY OUTCOMES:
Cost-effectiveness | 1 year follow up
  cost-effectiveness will be measured with incremental cost-effectiveness ratio (ICER)